CLINICAL TRIAL: NCT04155749
Title: Master Protocol for the Phase 1 Study of Cell Therapies for the Treatment of Patients With Relapsed Refractory Multiple Myeloma, Including Long-term Safety Follow-up
Brief Title: Study of Anitocabtagene-autoleucel in Participants With Relapsed Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Collaborators: Arcellx, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC-101-ARM1
Record Dates: First submitted 2019-10-17; First posted 2019-11-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Relapsed and Refractory Multiple Myeloma
Keywords: BCMA; Myeloma; Chimeric
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARM 1 (Experimental): Phase I study of BCMA-specific CAR-modified T-cell therapy using alternative binding domain, for the treatment of patients with relapsed and refractory multiple myeloma
  Interventions: Drug: anitocabtagene-autoleucel

INTERVENTIONS:
Drug: anitocabtagene-autoleucel — Chimeric Antigen Receptor T cells

SUMMARY:
Master protocol for cell therapy, Phase 1 proof-of-concept studies in relapsed and refractory multiple myeloma and includes long-term safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed and refractory Multiple Myeloma treated with at least 3 prior regimens of system therapy including Proteosome Inhibitor (PI), immunomodulatory drugs (IMiD), and anti-CD38 antibody (CD38mab); or has "triple-refractory" disease
* Documented measurable disease
* Adequate organ function
* Life expectancy > 12 weeks, Eastern Cooperative Group Performance Status 0-1

Exclusion Criteria:

* Plasma Cell Leukemia or History of Plasma Cell Leukemia
* Patients with a history of severe hypersensitivity to DMSO should be excluded
* Contraindication to fludarabine or cyclophosphamide
* Severe uncontrolled intercurrent illness (e.g., infection) or laboratory abnormalities
* Active central nervous system disease involvement by malignancy or active CNS pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), including DLT(s) | 24 months
Establish the RP2D of the investigational agent | 24 months

SECONDARY OUTCOMES:
Best overall response (BOR) by International Myeloma Working Group (IMWG) Consensus Criteria | 24 months
Overall Response Rate (ORR) by IMWG Consensus Criteria | 24 months
PK Parameter for Anitocabtagene-Autoleucel: Cmax | Day 1 up to 24 months
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter for Anitocabtagene-autoleucel: Tmax | Day 1 up to 24 months
  Tmax is defined as the time (observed time point) of Cmax.
PK Parameter for Anitocabtagene-Autoleucel: Area under the curve (AUC) | Day 1 up to 24 months
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Arcellx, Inc., Study Director — Arcellx, Inc.
Locations (4):
- United States (4):
  - Advanced Cellular Therapeutics Facility, DCAM 0800A, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buonato JM, Edwards JP, Zaritskaya L, Witter AR, Gupta A, LaFleur DW, Tice DA, Richman LK, Hilbert DM. Preclinical Efficacy of BCMA-Directed CAR T Cells Incorporating a Novel D Domain Antigen Recognition Domain. Mol Cancer Ther. 2022 Jul 5;21(7):1171-1183. doi: 10.1158/1535-7163.MCT-21-0552. PMID 35737298
- [Derived] Frigault MJ, Bishop MR, Rosenblatt J, O'Donnell EK, Raje N, Cook D, Yee AJ, Logan E, Avigan DE, Jakubowiak A, Shaw K, Daley H, Nikiforow S, Griffin F, Cornwell C, Shen A, Heery C, Maus MV. Phase 1 study of CART-ddBCMA for the treatment of subjects with relapsed and refractory multiple myeloma. Blood Adv. 2023 Mar 14;7(5):768-777. doi: 10.1182/bloodadvances.2022007210. PMID 35468618
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT04155749